CLINICAL TRIAL: NCT03611374
Title: Regional Anesthesia for Cardiothoracic Enhanced Recovery (RACER) for Patients Undergoing Sternotomy for Congenital Heart Repair
Brief Title: Regional Anesthesia for Cardiothoracic Enhanced Recovery (RACER) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Thomas Caruso, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 47032
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Congenital Heart Defect; Congenital Heart Disease; Anesthesia, Local; Opioid Use
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Erector Spinae Plane Block (Experimental): All participants will get the Erector Spinae Plane block (ESPB) as a prospective cohort study. After anesthesia induction all enrolled patients will have bilateral ESPB catheters placed at the T7 spine level prior to surgery. The surgery is a sternotomy for congenital heart repair in high risk children and adults.
  Interventions: Procedure: Bilateral Erector Spinae Plane Block (ESPB)

INTERVENTIONS:
Procedure: Bilateral Erector Spinae Plane Block (ESPB) — Bilateral ESPBs will be placed after anesthesia induction in eligible and consented patients who are undergoing a sternotomy for congenital heart repair. Patients will receive a local anesthetic agent through each catheter prior to surgery start. If possible, levels of the local anesthetic will be measured during the case. After surgery, patients will be admitted to the CVICU and extubation will be managed by the CVICU team. The ESPB group will have an automatic, alternating side boluses of the local anesthetic started through their nerve block catheters. Levels of the local anesthetic will be measured at intervals.

SUMMARY:
The erector spinae plane block is a novel regional anesthetic technique that allows for analgesia of the thorax and abdomen with a peripheral nerve block. The goals of this study are to determine if bilateral erector spinae plane blocks (ESPB) after sternotomy for congenital heart repair in high risk children and adults can decrease outcomes such as duration of postoperative mechanical ventilation (MV), perioperative opioid consumption, days in the intensive care unit (ICU) and length of stay (LOS).

ELIGIBILITY:
Inclusion Criteria:

i) Ages 0-99 ii) Give consent/parental consent to participate in study iii) Patients undergoing sternotomy for congenital heart repair surgeries

Exclusion Criteria:

i) Participants who do not consent or have parental consent ii) Patients who are clinically unstable or require urgent/emergent intervention iii) Patients under 5kg

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Median time to extubation in patients with ESPB | Duration of postoperative recovery (typically 1-2 weeks)
Median Cardiovascular Intensive Care Unit (CVICU) LOS in patients with ESPB | Duration of postoperative recovery (typically 1-2 weeks)
Determine average post-operative pain scores in patients with ESPB | Duration of postoperative recovery (typically 1-2 weeks)
Determine opioid consumption | Duration of postoperative recovery (typically 1-2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Caruso, MD, MEd, Principal Investigator — Stanford University
Locations (1):
- Lucile Packard Children's Hospital Stanford, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kain ZN, Fitch JC, Kirsch JR, Mets B, Pearl RG. Future of anesthesiology is perioperative medicine: a call for action. Anesthesiology. 2015 Jun;122(6):1192-5. doi: 10.1097/ALN.0000000000000680. No abstract available. PMID 25886775
- [Background] Ramamoorthy C, Haberkern CM, Bhananker SM, Domino KB, Posner KL, Campos JS, Morray JP. Anesthesia-related cardiac arrest in children with heart disease: data from the Pediatric Perioperative Cardiac Arrest (POCA) registry. Anesth Analg. 2010 May 1;110(5):1376-82. doi: 10.1213/ANE.0b013e3181c9f927. Epub 2010 Jan 26. PMID 20103543
- [Background] Fukunishi T, Oka N, Yoshii T, Kobayashi K, Inoue N, Horai T, Kitamura T, Okamoto H, Miyaji K. Early Extubation in the Operating Room after Congenital Open-Heart Surgery. Int Heart J. 2018 Jan 27;59(1):94-98. doi: 10.1536/ihj.16-630. Epub 2018 Jan 15. PMID 29332913
- [Background] Bhalla AK, Yehya N, Mack WJ, Wilson ML, Khemani RG, Newth CJL. The Association Between Inhaled Nitric Oxide Treatment and ICU Mortality and 28-Day Ventilator-Free Days in Pediatric Acute Respiratory Distress Syndrome. Crit Care Med. 2018 Nov;46(11):1803-1810. doi: 10.1097/CCM.0000000000003312. PMID 30028363
- [Background] Agarwal HS, Wolfram KB, Saville BR, Donahue BS, Bichell DP. Postoperative complications and association with outcomes in pediatric cardiac surgery. J Thorac Cardiovasc Surg. 2014 Aug;148(2):609-16.e1. doi: 10.1016/j.jtcvs.2013.10.031. Epub 2013 Nov 23. PMID 24280709
- [Background] Diaz LK. Anesthesia and postoperative analgesia in pediatric patients undergoing cardiac surgery. Paediatr Drugs. 2006;8(4):223-33. doi: 10.2165/00148581-200608040-00002. PMID 16898853
- [Background] Anand KJ, Hickey PR. Halothane-morphine compared with high-dose sufentanil for anesthesia and postoperative analgesia in neonatal cardiac surgery. N Engl J Med. 1992 Jan 2;326(1):1-9. doi: 10.1056/NEJM199201023260101. PMID 1530752
- [Background] Pollak U, Serraf A. Pediatric Cardiac Surgery and Pain Management: After 40 Years in the Desert, Have We Reached the Promised Land? World J Pediatr Congenit Heart Surg. 2018 May;9(3):315-325. doi: 10.1177/2150135118755977. PMID 29692232
- [Background] Brix-Christensen V. The systemic inflammatory response after cardiac surgery with cardiopulmonary bypass in children. Acta Anaesthesiol Scand. 2001 Jul;45(6):671-9. doi: 10.1034/j.1399-6576.2001.045006671.x. PMID 11421823
- [Background] Gaudilliere B, Fragiadakis GK, Bruggner RV, Nicolau M, Finck R, Tingle M, Silva J, Ganio EA, Yeh CG, Maloney WJ, Huddleston JI, Goodman SB, Davis MM, Bendall SC, Fantl WJ, Angst MS, Nolan GP. Clinical recovery from surgery correlates with single-cell immune signatures. Sci Transl Med. 2014 Sep 24;6(255):255ra131. doi: 10.1126/scitranslmed.3009701. PMID 25253674
- [Background] Fragiadakis GK, Gaudilliere B, Ganio EA, Aghaeepour N, Tingle M, Nolan GP, Angst MS. Patient-specific Immune States before Surgery Are Strong Correlates of Surgical Recovery. Anesthesiology. 2015 Dec;123(6):1241-55. doi: 10.1097/ALN.0000000000000887. PMID 26655308
- [Background] Hickey PR, Hansen DD. High-dose fentanyl reduces intraoperative ventricular fibrillation in neonates with hypoplastic left heart syndrome. J Clin Anesth. 1991 Jul-Aug;3(4):295-300. doi: 10.1016/0952-8180(91)90223-a. PMID 1910797
- [Background] Chaudhary V, Chauhan S, Choudhury M, Kiran U, Vasdev S, Talwar S. Parasternal intercostal block with ropivacaine for postoperative analgesia in pediatric patients undergoing cardiac surgery: a double-blind, randomized, controlled study. J Cardiothorac Vasc Anesth. 2012 Jun;26(3):439-42. doi: 10.1053/j.jvca.2011.10.012. Epub 2011 Dec 16. PMID 22176767
- [Background] Olivier JF, Bracco D, Nguyen P, Le N, Noiseux N, Hemmerling T; Perioperative Cardiac Surgery Research Group (PeriCARG). A novel approach for pain management in cardiac surgery via median sternotomy: bilateral single-shot paravertebral blocks. Heart Surg Forum. 2007;10(5):E357-62. doi: 10.1532/HSF98.20071082. PMID 17855198
- [Background] Chakravarthy M, Thimmangowda P, Krishnamurthy J, Nadiminti S, Jawali V. Thoracic epidural anesthesia in cardiac surgical patients: a prospective audit of 2,113 cases. J Cardiothorac Vasc Anesth. 2005 Feb;19(1):44-8. doi: 10.1053/j.jvca.2004.11.008. PMID 15747268
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Kose HC, Kose SG, Thomas DT. Lumbar versus thoracic erector spinae plane block: Similar nomenclature, different mechanism of action. J Clin Anesth. 2018 Aug;48:1. doi: 10.1016/j.jclinane.2018.03.026. Epub 2018 Apr 9. No abstract available. PMID 29649625
- [Background] Tsui BCH, Navaratnam M, Boltz G, Maeda K, Caruso TJ. Bilateral automatized intermittent bolus erector spinae plane analgesic blocks for sternotomy in a cardiac patient who underwent cardiopulmonary bypass: A new era of Cardiac Regional Anesthesia. J Clin Anesth. 2018 Aug;48:9-10. doi: 10.1016/j.jclinane.2018.04.005. Epub 2018 May 26. No abstract available. PMID 29684728